CLINICAL TRIAL: NCT03522207
Title: Stabilisation de la qualité du Sommeil Chez le Sujet en Douleurs Orofaciales Chroniques - étude expérimentale en chassé croisé : Trazodone/ Placebo
Brief Title: Accuracy and Efficacy of Trazodone (Desyrel) on Sleep Quality and Pain Management of TMD Patient
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: shortstaff at sleep lab
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17.322
Record Dates: First submitted 2018-04-16; First posted 2018-05-11 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: TMD; Sleep Bruxism; TMJ Pain; Chronic Pain; Sleep Disorder
MeSH Terms: conditions — Sleep Bruxism; Chronic Pain; Sleep Wake Disorders | interventions — Polysomnography; Trazodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trazo1 (Experimental): After a baseline polysomnography (PSG), subject will receive 100 mg of trazodone 30 minutes prior to their 2nd PSG and will receive 100mg Placebo 30 minutes prior to their 3rd PSG.
  Interventions: Diagnostic Test: polysomnography; Drug: Trazodone; Drug: placebos
- Trazo2 (Experimental): After a baseline polysomnography (PSG), subject will receive 100 mg of placebo 30 minutes prior to their 2nd PSG and will receive 100mg trazodone 30 minutes prior to their 3rd PSG.
  Interventions: Diagnostic Test: polysomnography; Drug: Placebos; Drug: Trazodone

INTERVENTIONS:
Diagnostic Test: polysomnography — BASELINE PSG Patient has to sleep over at the hospital (sleep lab). The technician will place several sensors on your scalp, temples, chest and legs to record all the data needed for your evaluation. You will be monitored throughout the duration of the test (approximately 6 hours). Brain waves, eye movements, chin muscle tone, breathing patterns, snoring, heart rate, blood pressure, blood oxygen level, body position and muscle activity will be recorded.
Drug: Trazodone — 100 mg trazodone or placebo given once 30 minutes prior to 2nd PSG
  Arms: Trazo1
Drug: Placebos — placebo per os 30 minutes prior to 2nd PSG
  Arms: Trazo2
Diagnostic Test: polysomnography — 2nd psg, done 1 week after baseline. Patient has to sleep over at the hospital (sleep lab). The technician will place several sensors on your scalp, temples, chest and legs to record all the data needed for your evaluation. You will be monitored throughout the duration of the test (approximately 6 hours). Brain waves, eye movements, chin muscle tone, breathing patterns, snoring, heart rate, blood pressure, blood oxygen level, body position and muscle activity will be recorded.
Drug: Trazodone — 100 mg trazodone per os 30 minutes prior to 3rd PSG
  Arms: Trazo2
Drug: placebos — 100 mg placebo per os 30 minutes prior to 3rd PSG
  Arms: Trazo1
Diagnostic Test: polysomnography — 3rd PSG, done 2 weeks after baseline. Patient has to sleep over at the hospital (sleep lab). The technician will place several sensors on your scalp, temples, chest and legs to record all the data needed for your evaluation. You will be monitored throughout the duration of the test (approximately 6 hours). Brain waves, eye movements, chin muscle tone, breathing patterns, snoring, heart rate, blood pressure, blood oxygen level, body position and muscle activity will be recorded.

SUMMARY:
The objective is to evaluate the accuracy and efficacity of 1 dose of trazodone in TMD patient (with chronic orofacial pain and poor sleep quality).

Subject will have 3 polysomnography (PSG) over 3 weeks. The first one being the baseline.

Half of the patient will receive trazodone on their 2nd PSG and placebo on their 3rd PSG, and the other half will receive placebo bedofe their 2nd PSG and trazodone for the 3rd PSG.

Pain quality and sleep quality will be assessed before and after PSG. polysomnograms from baseline, placebo night and trazodone night will also be compared.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) is an umbrella term to describe different disorders that affect the temporomandibular joint (TMJ) and/or muscles of mastication 1. TMD is one of the most common chronic orofacial pain conditions and the second most commonly occurring musculoskeletal condition, affecting 5-12% of the U.S and Canada. As other chronic pain conditions, TMD significantly impacts patients' quality of life (sleep quality, mood, eating, energy, etc). It is frequently associated with psychological conditions such as anxiety, depression, or somatization, which are often related with central sensitization and disability. The importance of the psychological axis for diagnose and treat TMD along with other orofacial pain disorders is reflected in the ongoing process of including psychosocial variables in the new orofacial pain classification.

The NIH funded Orofacial Pain Prospective Evaluation and Risk Assessment (OPPERA) study is probably one of the most important and well-funded investigations assessing risk factors for new onset and chronicity of TMD. This comprehensive study found that other comorbidities, self-report of jaw parafunction, and somatization were important predictors for clinical TMD. It was also found that deteriorated subjective sleep quality, assessed using the Pittsburgh Sleep quality Index (PSQI), it is present in TMD patients, can also predict incidence of TMD.

Sleep quality can be assessed subjectively or objectively:

1. Subjectively, it has been defined as tiredness on waking and throughout the day, feeling rested and restored on waking, and the number of awakenings they experienced in the night. It is usually assessed by self-report through questionnaires, such as the PSQI or visual analogue or category scales. Numerous studies, see above, reported poor subjective sleep quality in TMD subjects; a finding that has also been observed in different chronic pain conditions such as fibromyalgia or neuropathic pain.
2. Objectively, sleep quality is assessed through polysomnographic evaluation (PSG), and it is defined as sufficient duration (> 7hrs), high efficiency (> 85%), and low fragmentation (< 25), as well as proper staging of sleep. Smith et al showed that sleep disturbances and sleep disorders are prevalent among TMD patients using PSG; and Dubrovsky et al. compared sleep architecture of 126 TMD cases with 46 matched controls, finding that in TMD patients there was an increase of N1 stage of sleep, an increase in arousals associated with respiratory events, and also in respiratory effort related arousals (RERAs).

Therefore, the results of these studies suggest that patients with TMD present decreased subjective and objective sleep quality when compared to controls.

The management of TMD frequently involves a multidisciplinary approach consisting on:

* Self-care measures with or without cognitive behavioral therapy (CBT).
* Physical therapy.
* Health psychology.
* Use of oral devices
* Short-term pharmacotherapy.

TMD is often accompanied by different medical comorbidities, including other pain disorders, psychological conditions, and sleep impairment, which complicate the clinical picture and make more difficult to manage it with usual strategies.

Thus, addressing the comorbid condition/status such as anxiety, depression, or poor sleep. becomes important for the success of the TMD treatment itself. In these cases, a therapy that can target symptomatology from different conditions seems like a beneficial approach for the complex TMD patient.

Cognitive behavioral therapy (CBT) and pharmacotherapy are two studied options for these cases. While CBT success is based on a long-term therapy, pharmacology can be beneficial for a short-term fast approach.

In TMD subjects, clonazepam, cyclobenzaprine, benzodiazepines, and tricyclic antidepressant have been studied with mixed-results in the improvement of sleep quality and pain. Evidence suggests that the antidepressant trazodone, a medication that is frequently prescribed off-label to manage insomnia, can help to attenuate the impact of sleep arousal in rising its thresholds in patients with obstructive sleep apnea (OSA). As a) TMD patients have been reported to present increased RERAs when compared to controls, b) OSA is a risk factor for TMD onset, c) OSA is present in about 1 out 3 subjects with TMD, and d) certain antidepressants have shown pain reduction properties , e) TMD is frequently associated psychological conditions that often interfere with sleep and chronify pain, Trazodone seems to be a putative candidate to improve sleep quality and pain in patients with TMD.

In normal subjects, Trazodone increases total sleep time and non-REM sleep duration without major side effects. Despite being an antidepressant, this medication is commonly prescribed to treat chronic and acute insomnia, anxiety disorders, and it has also been used to treat pain chronic conditions such as fibromyalgia.

Its use to improve sleep in OSA or chronic pain patients is off label and empirical so far, with limited studies done in controlled conditions. Interestingly and also empirically, the doses used to reduce to impact of sleep arousal and sleep instability and also to improve sleep quality seem to be in the 25-100 mg range, taken at bed time for one to 4 nights per week.

One of the most common side effects of trazodone, which perhaps can explain the advantage-effect of trazodone on sleep quality, is sedation. Other reported side effects are gastrointestinal (vomiting, diarrhea, constipation), cardiovascular (orthostatic hypotension in elderly or people with heart problems and tachycardia), and less commonly dry mouth, dizziness, blurred vision, headache, or change in weight.

Primary Hypothesis: Trazodone will contribute to reduce the sleep instability associated to poor sleep in TMD subjects.

Secondary Hypotheses: Trazodone will contribute to improve subjective sleep quality and to decrease pain ratings in TMD subjects.

Method:

Subjects: 16 patients with chronic TMD (defined below), aged 18 to 45 years, and reporting poor sleep quality will be recruited at the Université de Montréal dental clinic, at the CHUM stomatology department, and based on referrals from physicians and dentists in the community.

Since TMD is three time more prevalent in the female population, and in order to reduce variability in a relatively small sample size, only females will be recruited.

Sample size: The sample size is based on a previous study whit similar outcomes and design in OSA patients. After the recruitment of 10 participants, an exploratory power analysis with a conventional alpha of 0.05 and a power level 0.80 will be performed.

Experimental design:

Design: A crossover, double blind design with a 7-day washout period will be used. Patients will be recorded in blocks of 1 night at a time for a total of 3 nights (night 1 for baseline-habituation to sleep lab), night 2 or 3 for medication or placebo administered in a random double-blind fashion).

In Experimental nights 2 or 3: drug trazodone per os 100 mg/placebo (cross over, double blind design) after a 1 week for washout from treatment sequence #1.

Subjects will complete psychosocial and demographic questionnaires before baseline-habituation night, including sleep quality, day time stress, anxiety, depression, quality of life, alcohol or coffee use, awareness of clenching or grinding, presence of comorbidities, using research questionnaires or numerical rating scales.

Sleep recording will start at 22h30 and patients will be awakened at 7h30.

Drug administration: Trazodone (Desyrel) will be given in a crossover order with placebo. The order of administration of the active medication (trazodone) and placebo will be reversed for half of the subjects. Trazodone and placebo will be prepared by a pharmacist in identical size and color to maintain the blind conditions. Randomization will be done by the research pharmacy, and the randomization key will also be held the research pharmacy.

A dose of 100mg given at bedtime was elected since it was the dose used in the prior studies that showed increased thresholds arousals with no reported side effects.

Trazodone is absorbed within 30-60 min, with a maximum plasma level reached in 2-4 hours and a mean half-life of 12 hours.

Sleep recording variables:

Each subject will be studied for 3 consecutive nights:

1. the first will be to screen for associated conditions (such as sleep apnea [>5/hr of sleep], periodic limb movement [>10/hr], REM sleep behavior disorder, epileptic activity) and for adaptation to the sleep laboratory conditions. All recording will take place in a light and sound-attenuated room.
2. nights 2 and 3 will be the experimental nights.

During these nights, the following parameters will be recorded using surface electrodes: central and occipital EEG leads (C3A2; 02A1), right and left EOG, chin EMG, EMG from right and left masseteric (for sleep bruxism), and anterior tibialis muscles (for periodic limb movement), and heart rate (ECG) derivation (for tachycardia). Airflow, respiratory movements and oxygen saturation - CO2 for hypercapnia will be monitored during the first night to rule out sleep apnea syndrome, and during following night 2 and 3. Psychomotor vigilance task (PVT) will be performed at baseline and two experimental nights the next morning upon awakening.

The sleep recordings will start at 22:30 (10:30pm) and will stop when the subject spontaneously awakes or at 07:30am. Self-reports of pain, sleep quality, and side effects will be collected on the morning after administration of medication/placebo and 7-10 days after intervention.

Sleep scoring, EEG and ECG analysis: sleep scoring will be performed off-line on a computer screen under blind conditions for all studies, sleep stages will be scored visually according to a standard method.

For more stable measures during sleep and to avoid confounding influences, subjects will be free of: 1) over to counter medications for 48 hrs before the study; 2) alcohol, coffee, tea, cola, any cigarette, etc. 12 hrs before the study. Subjects will also eat a light dinner 3 hrs before sleep and will relax in the sleep laboratory for at least 90 min before going to bed.

Statistics and design for analysis: Results will be analyzed under blind conditions. Sleep parameters (microarousal, K-alpha complexes, etc.) for each night (2 and 3) and questionnaires (e.g., stress and sleep quality) will be analyzed with:

1. parametric tests such as: a) t-test for between-group comparisons, ANOVA and repeated measures ANOVA followed by Tukey and contrasts for post-hoc comparisons when appropriate (SAS and Systat statistical softwares); b) iterative general least squares (IGLS) for across-night time effects, or canonical correlations for first 4 non-REM episodes;
2. nonparametric tests such as: chi-square, Mann-Whitney (for category data and/or when data distribution is not normal);
3. Correlations tests, such as Pearson or Spearman, where appropriate.

The investigator will obtain the informed consent from the patient by means of a dated and signed declaration of informed consent before any study related procedure is performed.

Data will be stored using an alpha-numerical code corresponding the the patient's identification. The code will be kept using an excel file, protected by a password only known by the study coordinator and the principal investigator.

Medical data relevant to this study will be stored and analysed while maintaining confidentiality. All data transferred to the CRF and any process derived from the CRF will be handled anonymously. That will ensure that the identity of the individual will be protected.

All CRF will be kept in a locked file cabinet, located in room 221-H. All data will be kept for 10 years.

All results publication (abstract, scientific publication, congress, symposium, etc) will be done as a group of patients.

Trazodone may be potentially beneficial for long-term treatment in cases of chronic OFP complaining of poor sleep quality and, eventually, chronic morning headache patients without sleep disordered breathing.

The drug is administered in the hospital under medical supervision and sleep recording are conduct under technical supervision. A physician is available on call for adverse effect (dizziness, nausea, hypotension, etc.) management. Investigators will be available on call during the study.

ELIGIBILITY:
Inclusion Criteria:

* painful TMD, defined as chronic myalgia (>6 months) with/without accompanying arthralgia per DC/TMD.
* Pain should have been present 15 days in the last month
* Pain of moderate to severe average intensity (at least 4 out 10 in a verbal numerical rating scale) in the last week.
* Poor sleep quality according to specific question of PSQI questionnaire (response of fairly bad or very bad sleep quality in the las month).

Exclusion Criteria:

* Presence of any dental or orofacial pain disorder not meeting the above definition.
* Use of other pharmacological treatment for TMD or sleep during duration of the study. Patients will be asked to discontinue any of those treatments before starting the study.
* Use of any psychotropic medication or drug known to influence sleep or pain such as amphetamines, benzodiazepines, anticonvulsants, neuroleptics, or antidepressants.
* Alcohol or substance abuse.
* Presence of major neurological or psychiatric disorders, such as epilepsy, schizophrenia or major depression; other sleep disorders such as narcolepsy, sleep apnea syndrome (SAS) or REM sleep behavior disorder.
* Presence of cardiovascular or bleeding disorders.
* History of tachycardia.
* Contraindications to Trazodone: previous allergic reaction to Trazodone, patients taking MAOIs.
* Pregnancy or lactation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Sleep stability score | 8 hours after medication intake
  Based on visual analysis of these parameters:
  Sleep stage shifts: change from deeper to lighter sleep stage (stage 2, 3&4, REM toward stages 1 or 2); measured as number/hour.
  Awakening: presence of alpha and beta electroencephalography (EEG) activities, with rise in submental/chin muscle tone, lasting>10s; measured as number/hour.
  Movement arousal: an EEG pattern or awakening associated with major body movement; measured as number/hour.
  Microarousal (MA): abrupt shift in EEG frequency lasting more than 3s and less than 10, excluding spindles and K-complexes; measured as number/hour.
  Heart rate rapid fluctuations: acceleration of heart beat within 15s recorded by 2 electrodes at thoracic positions. Measured as number/hour.
  Presence and severity of abnormal values will be determined based on AASM recommended cutoffs. For value reference in TMD women participants, see Dubrovksy et al 2014. We hypothesize all these parameters would decrease in Trazodone group.

SECONDARY OUTCOMES:
Sleep quality score | 8 hours after medication intake
  Based on visual analysis of these parameters:
  Sleep duration: from time in bed to wake as estimated by EEG (minutes) Sleep efficiency: % time asleep/time in bed (time in minutes) Sleep fragmentation: index of all above criteria (point 1) number/hour Sleep latency: from light off to first sign of sleep on EEG (minutes). REM sleep latency: from sleep onset (on EEG) to first REM sleep stage (minutes).
  Presence and severity of abnormal values will be determined based on AASM recommended cutoffs. For references of values in TMD women participants, see Dubrovksy et al 2014. We hypothesize that sleep duration and efficiency will improve in Trazodone group, while sleep fragmentation, sleep latency, and REM sleep latency will decrease.

OTHER OUTCOMES:
Subjective sleep quality | 8 hours after medication intake
  Measured with a numerical rating scale (0 to 10) were 0 is poorest possible sleep quality and 10 is the greatest possible sleep quality
Clinical pain intensity | 8 hours after medication intake
  Measured with a numerical rating scale (0 to 100) were 0 is no pain and 100 is the most intense pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lavigne, Study Director — Université de Montréal
Locations (1):
- CHUM, Montreal, Quebec, Canada